CLINICAL TRIAL: NCT04038970
Title: A Phase II, Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of KN019 in Patients With Active Rheumatoid Arthritis While Receiving Methotrexate
Brief Title: Efficacy and Safety Study of KN019 in Rheumatoid Arthritis Patients With an Inadequate Response to Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KN019-201
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KN019 5mg/kg (Experimental): Intravenous (IV) solution, 5 mg/kg, Day 1, Day 15, Day 29; every 28 days thereafter, 12 months
  Interventions: Biological: KN019, 5mg/kg; Combination Product: Methotrexate
- KN019 10mg/kg (Experimental): Intravenous (IV) solution, 10 mg/kg, Day 1, Day 15, Day 29; every 28 days thereafter, 12 months
  Interventions: Biological: KN019, 10 mg/kg; Combination Product: Methotrexate
- Placebo (Placebo Comparator): Intravenous (IV) solution, Day 1, Day 15, Day 29; every 28 days thereafter, 12 months
  Interventions: Biological: Placebo; Combination Product: Methotrexate

INTERVENTIONS:
Biological: KN019, 5mg/kg — Solution, intravenous, 5 mg/kg
  Arms: KN019 5mg/kg
Biological: KN019, 10 mg/kg — Solution, intravenous, 10 mg/kg
  Arms: KN019 10mg/kg
Biological: Placebo — Solution, intravenous, Placebo
  Arms: Placebo
Combination Product: Methotrexate — Tablets, oral, 7.5-25 mg weekly to be adjusted according to patient condition

SUMMARY:
The purpose of this study is to assess the efficacy, pharmacokinetics, safety, and immunogenicity of KN019 after intravenous administration on background methotrexate in patients with active rheumatoid arthritis and inadequate response to methotrexate.

DETAILED DESCRIPTION:
This study is designed to provide efficacy data in support of the proposed claims of reducing signs and symptoms, improvement in physical function, and 1 year safety data for KN019 dosed at 5 and 10 mg/kg in patients with inadequate response to stable weekly doses of background methotrexate.

ELIGIBILITY:
Key Inclusion Criteria:

* The patient must meet the American College of Rheumatology (ACR) classification criteria for the diagnosis of rheumatoid arthritis (RA) by satisfying at least four of the seven criteria;
* Patients must have been taking methotrexate for at least 3 months with at least a weekly dose of 7.5-25 mg, and a stable dose for 28 days prior to treatment (Day 1)
* The patient must have active disease at both screening and baseline, as defined by having both:

  6 tender/painful joints on motion (out of 68 joints assessed); and; 6 swollen joints (out of 66 joints assessed); CRP ≥ 7 mg/L, or ESR ≥28 mm/h

Key Exclusion Criteria:

* Pregnant or lactating females.
* History of any other autoimmune rheumatic disease.
* Patients who have previously received CTLA4-Ig therapy for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants the proportion of subjects meeting the American College of Rheumatology criteria for 20% improvement (ACR 20) on Day 169 | At Day 169
  The ACR 20 is based on 20% improvement (compared with baseline values) in tender and swollen joint counts and on 20% improvement in 3 of the remaining 5 core set measures (participant global assessment of pain, participant global assessment of disease activity, physician global assessment of disease activity, participant assessment of physical function) and 1 acute phase reactant value.

CONTACTS AND LOCATIONS:
Locations (1):
- Pingxiang people's hospital, Pingxiang, Pingxiang, China